CLINICAL TRIAL: NCT04901832
Title: Effectiveness of Intradialytic Stretching Exercises on Prevention and Reduction of Leg Muscle Cramps Among Patients Undergoing Hemodialysis: Randomized Controlled Trial
Brief Title: Intradialytic Stretching Exercises on Prevention and Reduction of Leg Muscle Cramps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kufa University (Other)
Responsible Party: Principal Investigator, Amjed Abdulabbas Shraida, Principal Investigator, Kufa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IDSE-1
Record Dates: First submitted 2021-05-19; First posted 2021-05-26 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Muscle Cramp
Keywords: Stretching Exercises, Muscle Cramps, Hemodialysis.
MeSH Terms: conditions — Muscle Cramp

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The intervention in this group is stretching exercises with the aim of prevention and reduction of leg muscle cramps among patients undergoing hemodialysis
  Interventions: Other: Intradialytic stretching exercises
- Control Group (No Intervention): The participants in this group used as reference group

INTERVENTIONS:
Other: Intradialytic stretching exercises — Exercises performed actively and passively to reduce or prevent muscle cramps during hemodialysis procedure.
  Arms: Experimental Group

SUMMARY:
Renal replacement therapy is a treatment option for people who have acute or chronic renal failure. A patient with increasing symptoms of renal failure is referred to a dialysis and transplantation center early in the course of progressive kidney disease. Hemodialysis is one of the most widely used dialysis procedures. Muscle cramps are the most common complication experienced by hemodialysis patients that usually develop during and in between hemodialysis therapy. These cramps appear to be the most common reason for the early termination of the hemodialysis session.

- Research Question: Is there a difference in leg muscle cramps levels between patients undergoing hemodialysis who received intradialytic stretching exercises compared to those patients who do not receive these exercises?

- Hypothesis: Leg muscle cramp levels are less among patients undergoing hemodialysis who receive intradialytic stretching exercises compared to those patients who do not receive such exercises.

DETAILED DESCRIPTION:
Study Sample:

Non-probability purposive sample of 60 patients undergoing hemodialysis. The sample is divided randomly into two groups; 30 patients as study group are exposed to intradialytic stretching exercises, and the other 30 patients are not exposed to the exercises considered as the control group.

The Study Instrument:

To determine the effectiveness of the intradialytic stretching exercises program on the prevention and reduction of leg muscle cramps among patients undergoing hemodialysis, the researcher has adopted an assessment tool in order to achieve each of the study objectives. This tool consists of three parts:

Part I: Socio-Demographic Data:

A socio-demographic datasheet consists of (6) items, which include residency, gender, age, smoking, educational level, occupational status. These variables are coded as preparation for data analysis.

Part II: Clinical Variable:

The second part of the questionnaire consists of (10) items, which include duration of dialysis treatment, number of hemodialysis session per week, duration of hemodialysis session, frequency of leg muscle cramps per week, site of leg muscle cramps, comorbidity, level of calcium, body mass index, ultrafiltration rate, and ultrafiltration volume. These variables are coded as preparation for data analysis.

Part III: Muscle Cramp questionnaire chart. The muscle cramp questionnaire chart is adopted to assess the level of muscle cramps during hemodialysis, before and after the intervention. This chart is used because it is an easy and valid tool, as it has been adopted in several previous studies. It contains various features of muscle cramps such as the frequency of muscle cramps, duration of muscle cramps, level of pain, temperature, and discomfort which was comprehensively scored as the level of muscle cramps ranging from (0-13).

Score Interpretation of Study Instruments :

Four scores are used for rating the levels of leg muscle cramps among Patients undergoing Hemodialysis in terms of no cramps, mild cramps, moderate cramps, and severe cramps. These cramps levels are scored as (0) for no cramps, (1 - 4) for Mild cramps, (5 - 8) for moderate cramps, and (9 - 13) for severe cramps.

Regarding the body mass index, four scores are used for rating the body mass index categories in terms of underweight, normal, overweight, obesity. These categories are scored as shown in the following table from Centers for Disease Control and Prevention, (2020) Underweight:Below 18.5 Normal or Healthy Weight:18.5 - 24.9 Overweight:25.0 - 29.9 Obese:30.0 and Above

Data collection The Data Collection was done according to CONSORT 2010 Flow Diagram

ELIGIBILITY:
Inclusion Criteria:

* Patients with age group 20-60 years, because it is the most common age group affected by CKD and they appropriate to apply for the study program.
* Both male and female patients who are undergoing hemodialysis and suffer from muscle cramps.
* Patients who are receiving two or more HD sessions a week, to facilitate patients follow-up.
* Patients who are willing to participate, because the patients' participation is voluntary.
* Patients who are alert and able to communicate verbally, to make the program applicable and facilitate the data collection.

Exclusion Criteria:

* Emergency hemodialysis patients, to avoid mal-efficient (harmlessly apply the program).
* Patients with vascular access in a lower extremity, to avoid vascular access failure.
* Patients with skin sores, wounds, dermatitis, or edema of the lower extremities, with a known history of deep vein thrombosis (DVT), peripheral vascular disease (PVD), or peripheral neuropathy, to prevent complications.
* Patients who are unable to communicate, because the patients' communication is an essential part of data collection.
* Patients who suffer from breathing difficulty, because the application of the program required patients compliance and may cause fatigue among involved patients
* Not willing to participate, because the patients' participation is voluntary.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-13 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
Muscle cramp questionnaire chart | 4 week muscle cramp assessment
  The muscle cramp questionnaire chart is adopted to assess the level of muscle cramps during hemodialysis, before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Diaa K Abd-Ali, Dr., Study Director — University of Al-Ameed. College of Nursing
Locations (1):
- Al-Sadder Medical City / The Specialized Center for Kidney Diseases and Transplantation / Hemodialysis Unit, Kufa, Al Najaf, Iraq

IPD SHARING:
Plan to Share IPD: Yes
Any data that does not violate ethical considerations will be obtained from the researcher.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting in October 2021
Access Criteria: Researchers in medical colleges (bachelors, masters, and doctorates), the Iraqi Ministry of Higher Education and Research, and the Iraqi Ministry of Health can access the data by emailing the researcher.